CLINICAL TRIAL: NCT00225303
Title: A Phase II, Randomized, Active Controlled, Open Label Trial to Investigate the Efficacy and Tolerability of TMC125 in HIV-1 Infected Subjects, Who Are PI-na�ve and With Documented Genotypic Evidence of NNRTI Resistance From Previous NNRTI Use.
Brief Title: TMC125-C227: A Phase II Randomized, Active-Controlled, Open Label Trial to Investigate the Efficacy and Tolerability of TMC125 in HIV-1 Infected Subjects, Who Are PI-Naive and With Documented Genotypic Evidence of NNRTI Resistance From Previous NNRTI Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006730
Record Dates: First submitted 2005-09-12; First posted 2005-09-23 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection
Keywords: HIV infection; TMC125; Non-Nucleoside reverse transcriptase inhibitor; Protease inhibitor; TMC125-C227
MeSH Terms: conditions — HIV Infections | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
The purpose of this study is to determinate the effectiveness, safety and tolerability (how well the body accepts the drug) of an investigational Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) called TMC125.

DETAILED DESCRIPTION:
Patients who have previously received a first HIV NNRTI containing regimen or who have received an NNRTI containing treatment for prevention of mother to child transmission (MTCT), and who have never used a protease inhibitor (PI) may be eligible to participate. TMC125 (at 800 mg b.i.d. of the old formulation and after the formulation switch, 200 mg b.i.d. of the new formulation) will be studied versus an active control (investigator selected PI). All patients will receive an underlying therapy containing 2 investigator selected NRTIs. 300 patients will be enrolled in Argentina, Brazil, Mexico, Peru, Chile, Costa Rica, Russia, South-Africa, Spain, Thailand, UK, USA, Thailand, India and Malaysia. The duration of the study is 48 weeks with an optional extension for patients in the TMC125 treatment group until virologic failure or commercial availability of the drug. TMC125 at 800mg twice daily of the old formulation; after the formulation switch, TMC125 at 200mg twice daily of the new formulation. The initial duration is 48 weeks with an optional extension for patients in the TMC125 treatment group until virologic failure or commercially availability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Documented HIV-1 infection
* Stable NNRTI-containing ART (minimum 12 weeks) at screening OR treatment interruption (minimum 4 weeks) at screening OR having received an NNRTI alone or in combination with other ARVs for prevention of MTCT
* Plasma viral load at screening above 1000 HIV-1 RNA copies/ml
* Prior NNRTI-experience with documented genotypic evidence of resistance to currently available NNRTIs (defined as at least one NNRTI-associated mutation per IAS-USA Drug resistance Mutation guidelines)
* Sensitive to the 2 NRTIs to be used as underlaying ART
* Subject has given informed consent

Exclusion Criteria:

* Previous treatment with Protease Inhibitors
* Presence of any currently active AIDS defining illness except stable cutaneous Kaposi's Sarcoma and Wasting syndrome due to HIV infection
* Current or past history of alcohol and/or drug use which, in the investigator's opinion, would compromise the subject's safety or compliance to the study protocol procedures
* Acute Hepatitis A, B or C or chronic hepatitis B or C with elevated LFTs of > 3 times ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Evaluate antiviral activity of TMC125 800mg twice daily and after the formulation switch, 200mg twice daily as part of an ART containing 2 NRTIs, by evaluating the proportion of subjects with plasma HIV-1 RNA levels < 50 copies/mL at 24 weeks.

SECONDARY OUTCOMES:
Evaluate: Antiviral activity, safety, tolerability and immunologic changes over treatment period with TMC125; Changes in viral genotype and drug susceptibility during trial; Efficacy, safety and tolerability of TMC125 compared with active control group.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Result] Ruxrungtham K, Pedro RJ, Latiff GH, Conradie F, Domingo P, Lupo S, Pumpradit W, Vingerhoets JH, Peeters M, Peeters I, Kakuda TN, De Smedt G, Woodfall B; TMC125-C227 study group. Impact of reverse transcriptase resistance on the efficacy of TMC125 (etravirine) with two nucleoside reverse transcriptase inhibitors in protease inhibitor-naive, nonnucleoside reverse transcriptase inhibitor-experienced patients: study TMC125-C227. HIV Med. 2008 Nov;9(10):883-96. doi: 10.1111/j.1468-1293.2008.00644.x. Epub 2008 Sep 14. PMID 18795960
- See also: A Phase II, randomized, active controlled, open label trial to investigate the efficacy and tolerability of TMC125 in HIV-1 infected subjects, who are PI-na�ve and with documented genotypic evidence of NNRTI resistance from previous NNRTI use. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=993&filename=CR006730_CSR.pdf